CLINICAL TRIAL: NCT05889520
Title: ASSESSMENT OF THE PRESENCE OF DERIVATIVES OF ULTRA-PROCESSED FOODS IN BREAST MILK- The UFIM (Ultraprocessed Foods In Breast Milk) Project
Brief Title: The UFIM (Ultraprocessed Foods In Breast Milk) Project
Acronym: UFIM
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Medical Doctor, Doctor of Philosophy, Full Professor, Federico II University
Other Study IDs: 163/2023
Record Dates: First submitted 2023-05-26; First posted 2023-06-05 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Child Malnutrition; Child Allergy; Maternal Exposure
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lactacting women who are breastfeeding full-term infants: Caucasian women aged between 18 and 35 who are breastfeeding full-term infants observed at Pediatrics Section of Department of Translational Medical Sciences (University of Naples Federico II)

SUMMARY:
In last decades, a change in dietary habits has been observed in industrialized countries characterized by a drastic increase in the consumption of ultra-processed foods (UPF, Ultra-Processed Foods). As defined by the NOVA classification, UPFs are industrial formulations of food substances added with colourings, flavourings, emulsifiers, thickeners and other additives. Among the main compounds of UPFs are the advanced glycation end-products (AGEs). Increasing evidence suggests an association between dietary exposure to AGEs and the development of chronic non-communicable diseases, such as obesity and allergies, in the general population, through increased oxidative stress and inflammation. Preliminary evidence suggests that a maternal diet rich in AGEs during pregnancy and lactation could negatively influence the composition of breast milk and have a negative impact on the infants health. However, data regarding the presence of derivatives of UPFs in breast milk are not available. The UFIM (Ultraprocessed Foods In Breast Milk) study aims at evaluate the presence of UPFs-derivatives compounds in breast milk.

ELIGIBILITY:
Inclusion Criteria:

Caucasian women who are breastfeeding full-term infants

Exclusion Criteria:

* Non-Caucasian ethnicity;
* Age <18 and >35 years;
* Mothers of preterm children;
* Non-exclusive breastfeeding;
* Mothers suffering from chronic, malignancies, immunodeficiencies, chronic infections, autoimmune, inflammatory bowel disease, celiac disease, genetic-metabolic diseases, cystic fibrosis and other chronic lung diseases, cardiovascular / respiratory / intestinal malformations, neuropsychiatric disorders and pathologies neurological, vegetarian and vegan diet;
* Mothers with tattoos, scars, moles or skin lesions on both forearms.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Caucasian women aged between 18 and 35 who are breastfeeding full-term infants observed at Pediatrics Section of Department of Translational Medical Sciences (University of Naples Federico II)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
To evaluate the presence of the major UPFs-derived compounds AGEs in breast milk | 36 months
  Through the liquid chromatography with triple quadrupole mass spectrometric detection techniques (LC-MS/MS) will be assessed the quantity of AGEs in breast milk.

SECONDARY OUTCOMES:
Dietary intake of UPF in lactating women | 36 months
  A 7-day food diary will be used for the evaluation of UPF dietary intake through the NOVA classification system.
Dietary intake of AGEs in lactating women | 36 months
  A 7-day food diary will be used for the evaluation of AGEs dietary intake through a reference database reporting the presence of AGEs in food.
Skin AGEs accumulation levels in lactating women | 36 months
  The non-invasive device AGEs reader will be used to evaluate the skin AGEs accumulation levels in lactating women.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No